CLINICAL TRIAL: NCT00646672
Title: Assessment of Cerebral Circulation and Perfusion in Adults After Neonatal Carotid Occlusion
Brief Title: Aneurysms and Carotid Artery Block in Newborns
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080095; 08-N-0095
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-04-16

CONDITIONS: Cerebrovascular Disorder
Keywords: ECMO; Cerebral Perfusion; Carotid Artery; Aneurysm; Cerebral Circulation; Common Carotid Artery Occlusion
MeSH Terms: conditions — Cerebrovascular Disorders; Aneurysm

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study will determine the risk of brain aneurysm (abnormal outpouching of a brain artery) in young adults who had their carotid artery tied off as an infant as part of the extracorporeal membrane oxygenation (ECMO) procedure. This procedure is sometimes performed on newborns with lung problems so that they can have oxygen brought to their blood outside the body. ECMO operates similar to a heart-lung machine. Blood drained from the veins has the carbon dioxide removed and oxygen added. The oxygenated blood is then returned to the body through the arteries.

People 18 to 25 years of age who underwent ECMO as an infant at the Children's National Medical Center in Washington, D.C., may be eligible for this study.

Participants undergo the following procedures:

* Medical history and physical and neurological examinations.
* Magnetic resonance imaging (MRI) of the head and neck. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The subject lies in the scanner (a metal cylinder surrounded by a magnetic field) for about 90 minutes, lying still for up to 15 minutes at a time. During part of the procedure, a contrast dye is injected into a vein through a catheter (thin plastic tube) to enhance the images.

DETAILED DESCRIPTION:
Objective:

To assess whether the hemodynamic stress of long-term common carotid artery occlusion can lead to cerebral aneurysm formation in young adults.

Study population:

100 adults 18-25 years of age who underwent common carotid artery (CCA) occlusion as a neonate as part of the extracorporeal membrane oxygenation (ECMO) procedure performed in the setting of pulmonary insufficiency.

Design:

Patients who underwent CCA occlusion as a neonate for ECMO at Children's National Medical Center will be identified and contacted. The study will be explained and informed consent will be obtained. Subjects will undergo outpatient evaluation to include history and physical, magnetic resonance angiography and magnetic resonance imaging of the head.

Outcome measures:

* Cerebrovascular anatomic anomalies such as cerebral aneurysms and persistent fetal circulation pathways, etc.
* Cerebral perfusion asymmetry on MRI.
* Cerebral parenchymal abnormalities such as stroke.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 18-25 years of age.

Subjects had VA ECMO as a neonate at Children's National Medical Center.

Subjects must be in good health.

Subjects must provide informed, written consent for participation in this study.

EXCLUSION CRITERIA:

Subjects with a history or evidence of mental retardation precluding a written consent unless this consent could be obtained from a legal guardian.

Subjects with a history of reaction to MR contrast media or who are unable to have an MRI.

Subjects who underwent carotid artery reconstruction after neonatal ECMO.

Females who are pregnant or nursing.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03-17; Study Completion 2010-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrews RJ, Spiegel PK. Intracranial aneurysms. Age, sex, blood pressure, and multiplicity in an unselected series of patients. J Neurosurg. 1979 Jul;51(1):27-32. doi: 10.3171/jns.1979.51.1.0027. PMID 448414
- [Background] Bartlett RH, Gazzaniga AB, Jefferies MR, Huxtable RF, Haiduc NJ, Fong SW. Extracorporeal membrane oxygenation (ECMO) cardiopulmonary support in infancy. Trans Am Soc Artif Intern Organs. 1976;22:80-93. PMID 951895
- [Background] Burt VL, Whelton P, Roccella EJ, Brown C, Cutler JA, Higgins M, Horan MJ, Labarthe D. Prevalence of hypertension in the US adult population. Results from the Third National Health and Nutrition Examination Survey, 1988-1991. Hypertension. 1995 Mar;25(3):305-13. doi: 10.1161/01.hyp.25.3.305. PMID 7875754